CLINICAL TRIAL: NCT06603402
Title: Low-Dose Involved-Field Radiotherapy Combined with Immunochemotherapy for Locally Advanced, Unresectable Esophageal Squamous Cell Carcinoma: a Prospective, Single-Arm, Phase II Study.
Brief Title: Low-Dose Involved-Field Radiotherapy Plus Immunochemotherapy for ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Clinical Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX-LION Study
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-09

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC); Immunotherapy
Keywords: Esophageal Squamous Cell Carcinoma; Radiotherapy; immunotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- low-dose involved-field radiotherapy combined with immunochemotherapy (Experimental): low-dose involved-field radiotherapy combined with immunochemotherapy
  Interventions: Radiation: low-dose involved-field radiotherapy combined with immunochemotherapy

INTERVENTIONS:
Radiation: low-dose involved-field radiotherapy combined with immunochemotherapy — low-dose involved-field radiotherapy combined with immunochemotherapy

SUMMARY:
The aim of this clinical trial is to evaluate whether low-dose involved-field radiotherapy combined with immunochemotherapy can reduce treatment-related adverse effects, enhance progression-free survival (PFS), and improve overall survival (OS) in patients with locally advanced, unresectable esophageal squamous cell carcinoma.

The key questions this study seeks to address are:

* Can low-dose involved-field radiotherapy combined with immunochemotherapy reduce treatment-related adverse effects?
* Does this combined approach improve PFS and OS in these patients?

Participants in the study will:

* Undergo an endoscopy at West China Hospital to confirm their diagnosis.
* Receive a treatment regimen that includes low-dose radiotherapy at 45.0 Gy in 1.8 Gy per fraction over 25 fractions, alongside immunochemotherapy, with three cycles of chemotherapy administered every 3 weeks.
* After completing the full treatment regimen, participants will undergo regular follow-up visits and monitoring by healthcare professionals.

DETAILED DESCRIPTION:
This is a single-arm, single-center, prospective clinical study aimed at evaluating the efficacy and safety of low-dose involved-field radiotherapy combined with immunochemotherapy in patients with locally advanced, unresectable esophageal squamous cell carcinoma (ESCC). The study will enroll subjects with pathologically confirmed ESCC (via histology or cytology), clinically staged as cT1-4aN+M0, who are deemed unsuitable for surgical intervention by the investigators or have declined surgical treatment.

Initially, patients will receive one cycle of induction immunochemotherapy consisting of paclitaxel or nab-paclitaxel plus carboplatin, in combination with camrelizumab administered at 200 mg intravenously every three weeks. On the first day of the second chemotherapy cycle, low-dose involved-field radiotherapy will commence. The radiotherapy protocol involves a total dose of 45.0 Gy delivered in 25 fractions of 1.8 Gy each (45.0 Gy/1.8 Gy per fraction over 25 fractions). The clinical target volume (CTV) is defined by extending the gross tumor volume (GTV) 3 cm superiorly and inferiorly, and 0.5 cm anteriorly, posteriorly, and laterally; for involved lymph nodes (GTVn), a 0.5 cm margin is added in all directions.

Following disease stabilization, patients will continue with maintenance therapy using camrelizumab monotherapy for up to one year or until disease progression, as assessed by RECIST 1.1 criteria, or the emergence of intolerable adverse effects. Upon completion of treatment, subjects will undergo routine follow-up according to standard care protocols to document survival status and long-term adverse reactions.

The study utilizes a historical control one-year progression-free survival (PFS) rate of 34% from definitive chemoradiotherapy in locally advanced ESCC. It is hypothesized that the combination of camrelizumab with dual-agent chemotherapy (paclitaxel or nab-paclitaxel plus carboplatin) and sequential low-dose involved-field radiotherapy will improve the 12-month PFS rate to 52%. Based on a two-sided significance level (α) of 0.05 and a power (1-β) of 80%, the required sample size is calculated to be 37 patients. Accounting for a 10% dropout rate, a total of 41 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Patients with locally advanced, unresectable ESCC who have received radical treatment (radical chemoradiotherapy or radical radiochemotherapy), including:

Cervical esophagus involvement, T4 stage, supraclavicular lymph node metastasis, or inability to tolerate or refusal of surgery due to personal reasons; Failure of neoadjuvant or conversion therapy;Unresectable local recurrence after surgery (with measurable target lesions)

* No evidence of tumor recurrence or metastasis on follow-up examination 2-3 weeks after radical treatment
* Ability to provide fresh tumor tissue specimens (baseline)
* Normal function of major organs
* Performance Status (PS) score ≤ 1
* Patients of childbearing potential must agree to use contraception.
* Voluntary participation with signed informed consent

Exclusion Criteria:

* History of fistula formation due to primary tumor invasion
* High risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation.
* Poor nutritional status
* Previous immune-related adverse events during prior radical treatment, including grade ≥3 immune-related pneumonitis, myocarditis, etc
* Presence of symptoms or signs of interstitial disease
* Patients with any severe and/or uncontrolled medical condition
* Presence of concurrent malignancies
* Presence of other autoimmune diseases or long-term use of immunosuppressants or corticosteroids.
* Patients who are difficult to communicate with or are unlikely to comply with long-term follow-up.
* Any other conditions that the investigator deems unsuitable for participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 41 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The safety of low-dose involved-field radiotherapy combined with immunochemotherapy | 12months
  This study will collected any adverse medical events that occurred during the study drug treatment, and the treatment-related adverse events as assessed by" CTCAE v5.0".

SECONDARY OUTCOMES:
The efficacy of low-dose involved-field radiotherapy combined with immunochemotherapy | 12months
  The 1-year Progression-free survival (PFS) rate will be evaluated as the primary endpoint using RECIST 1.1 criteria.
The efficacy of low-dose involved-field radiotherapy combined with immunochemotherapy | 12months
  Evaluate objective response rate (ORR) using the RECIST 1.1 criteria
The efficacy of low-dose involved-field radiotherapy combined with immunochemotherapy | 24months
  Using the RECIST1.1 tumor evaluation criteria for efficacy evaluation, evaluate overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: zhenyu ding, MD, Principal Investigator — West China Hospital, Sichuan University, China
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No